CLINICAL TRIAL: NCT06407440
Title: The Effect of Exercise Given to Cashiers Along With Ergonomics Training on Pain and Work Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Dr. Öğr. Üyesi Ömer Şevgin, Asst. Prof. Dr., Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uskudar7
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Work-related Illness; Work Related Upper Limb Disorder
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Active Comparator): Ergonomics training will be provided and followed up
  Interventions: Other: control
- exercise (Experimental): In addition to ergonomics training, exercise training will be provided.
  Interventions: Other: exercise

INTERVENTIONS:
Other: control — There will be no interference ergonomics training
  Arms: control
Other: exercise — upper extremity strengthening exercises upper extremity stretching exercises ergonomics training posture training relaxation exercises
  Arms: exercise

SUMMARY:
The aim of the study is to examine the effectiveness of the exercises given to cashiers through ergonomics training.

DETAILED DESCRIPTION:
The work will be done with 60 cashiers. These cashiers will be selected on the condition that they work at least 40 hours a week. 60 employees will be randomly divided into two groups of 30 people each. All participants will be given ergonomics training. In addition, participants in the exercise group will be given a 12-week exercise program. These two groups will be randomly divided into control and exercise groups. Each group will be evaluated twice, at the beginning and at the end of the study.

ELIGIBILITY:
inclusion criteria

* Those who have been working as cashiers in the market for at least 2 years
* Employees who have no obstacle to exercise
* Women and men aged 18-45
* Cashiers working 40 hours or more per week

exclusion criteria

* Being diagnosed with a serious psychological illness.
* Malignancy
* Advanced osteoporosis
* Being under 25 years of age.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-05-09 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2024-08-12 (Actual)

PRIMARY OUTCOMES:
Rapid Upper Limb Assessment | 14 weeks
  It is an ergonomics risk assessment method that quickly analyzes the employee's upper extremity from an ergonomic perspective. It evaluates upper extremity movements in 14 separate steps. 8 of these steps are scored for arm and hand position, and 6 for neck and trunk position, according to the table. The minimum Rapid Upper Limb Assessment Score = 1, and the maximum Rapid Upper Limb Assessment Score = 7. A high score means high risk.
occupational burnout scale | 14 weeks
  This scale aims to measure the degree of professional burnout that may occur due to stress in business life. It consists of 20 questions in total. For each question there are options: 'Never, Rarely, Sometimes, Often, Always'. The person will choose what suits him/herself.Possible score ranges for all scales is 0-100.Higher score is more favorable.
Nordic Extended Musculoskeletal Questionnaire | 14 weeks
  It is one of the questionnaires used to evaluate the severity and impact of musculoskeletal symptoms. In the survey, the frequency and severity of pain in the 'Neck, Shoulder, Upper Back, Elbow, Hand-wrist, Kala, Knee, Foot-ankle' areas of the body are evaluated in the last 12 months.It is a selection scale rather than a rating.
Pittsburgh Sleep Quality Index | 14 weeks
  This index evaluates sleep quality and disturbance over the past month. It contains a total of 24 questions. 19 of these questions are answered by the person's self-assessment, and 5 of them are answered by the roommate who shares the same room with the person. The 5 questions answered by the person's roommate are not included when calculating the score. In scoring, the lowest (0) and the highest (21) points are obtained. A score of 4 and above indicates poor sleep quality.
bournemouth neck survey | 14 weeks
  Since the Bournemouth Neck Pain Questionnaire evaluates individuals physically, mentally, emotionally and socially, it is a survey that can give an idea about the quality of life of individuals with chronic neck pain. In the survey, he evaluates the problems he has experienced in the last week in 7 questions. In scoring, the lowest is (0) and the highest is (70). As the score increases, pain intensity increases.

CONTACTS AND LOCATIONS:
Overall Officials: Devran YAŞAR, Study Chair — Uskudar University
Locations (1):
- Uskudar University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wasilewski RM, Mateo P, Sidorovsky P. Preventing work-related musculoskeletal disorders within supermarket cashiers: an ergonomic training program based on the theoretical framework of the PRECEDE-PROCEED model. Work. 2007;28(1):23-31. No abstract available. PMID 17264417
- [Background] Minghelli B, Ettro N, Simao J, Mauricio K. Work-related self-reported musculoskeletal disorders in hypermarket cashiers: a study in south of Portugal. Med Lav. 2019 Jun 28;110(3):191-201. doi: 10.23749/mdl.v110i3.7771. PMID 31268426
- [Background] Erick P, Sethatho M, Tumoyagae T, Letsholo B, Tapera R, Mbongwe B. Self-reported neck and back pain among supermarket cashiers in Gaborone, Botswana. Int J Occup Saf Ergon. 2023 Sep;29(3):989-997. doi: 10.1080/10803548.2022.2108653. Epub 2022 Sep 11. PMID 35930246
- [Background] Peter P, Elin J, Katarina K, Malin J. Differences in cashiers work technique regarding wrist movements when scanning groceries. Work. 2012;41 Suppl 1:5436-8. doi: 10.3233/WOR-2012-0845-5436. PMID 22317577
- [Background] Roxo LC, Ramos GC, Arruda ZM, Dias AC. Work activity and musculoskeletal symptoms in female cashiers. Rev Bras Med Trab. 2021 Sep 30;19(3):324-331. doi: 10.47626/1679-4435-2021-615. eCollection 2021 Jul-Sep. PMID 35774767
- [Derived] Yasar D, Safran EE, Sevgin O. The effect of combined ergonomic training and exercises on musculoskeletal pain and ergonomic risks in supermarket cashiers: a randomized controlled trial. Int Arch Occup Environ Health. 2025 Mar;98(2):255-265. doi: 10.1007/s00420-025-02132-z. Epub 2025 Mar 8. PMID 40056193